CLINICAL TRIAL: NCT01174251
Title: The Effect of General Anesthesia on the Risk for Arrhythmia -A Pilot Study
Brief Title: The Effect of General Anesthesia on the Risk for Arrhythmia
Acronym: 10-02725
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H61125-34760-01
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Arrhythmia
Keywords: general anesthesia; electrocardiography; long QT syndrome, acquired
MeSH Terms: conditions — Arrhythmias, Cardiac; Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Polymorphic ventricular tachycardia, known as Torsades de Pointes (TdP), is a specific form of ventricular arrhythmia with a characteristic twist of the QRS complex around the isoelectric baseline. TdP can degenerate into ventricular defibrillation followed by sudden cardiac death. A predictor for the development of TdP is the length of the QT interval measured on an EKG recording. The QT interval is known to be prolonged by many medications used in a perioperative setting as well as by other conditions such as hypothermia and electrolyte imbalance. General anesthesia exposes most of the investigators patients to a combination of several of those medications and conditions and therefore might increase the risk for the development of QT prolongation. Moreover, patient related risk factors are well known and aggravate the individual risk for potential life threatening TdP events when exposed to QT prolonging medications perioperatively.

Previous research suggests that more than 20% of the patients might develop QT prolongations perioperatively and are consequently on an increased risk for TdP; yet, no study has systematically investigated the magnitude of the problem and associated risk factors.

The proposed pilot study is designed as a prospective observational cohort study to investigate the QT interval before, during and after general anesthesia. It aims to determine the incidence of perioperative QT prolongations. A customary long term EKG recording device will be connected to a random sample of patients undergoing general anesthesia. Using these continuous EKG tracings, the lengths of the QT interval will be analyzed during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ASA I - III patients
* Age 18 years and older
* Scheduled for general anesthesia with a duration of at least 1 hour

Exclusion Criteria:

* Cardiac or thoracic surgery
* Planed postoperative ICU admission
* Non-English speaking
* Not in sinus rhythm
* Left and right bundle branch block
* Implanted pacemaker
* Mentally impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A simple random sample will be chosen among all patients scheduled for general anesthesia in the UCSF affiliations Mt. Zion Hospital and Moffit/Long Hospital meeting all inclusion- and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Kolodzie, M.D., PhD, Principal Investigator — Dept. of Anesthesia & Perioperative Care; University of California, San Francisco (UCSF)
Locations (1):
- UCSF Medical Center (Moffitt/Long, Mt. Zion), San Francisco, California, United States